CLINICAL TRIAL: NCT04707911
Title: Social Media Intervention to Stop Nicotine and Cannabis Vaping Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other); HopeLab Foundation (Other); Rescue Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T31IR1910; 21633 (Other: University of California, San Francisco); NCI-2021-11423 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Vaping
Keywords: Nicotine Dependence; Social Media
MeSH Terms: conditions — Vaping; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaping Intervention (Experimental): The vaping intervention will be implemented on Instagram. Participants in the treatment condition will be assigned to groups on Instagram, where they will receive up to 3 posts per day for 30 days. Groups are facilitated by a trained Guide, working with the Principal Investigator, Co-Investigators and a Pediatrician on demand if additional expertise or clinical advice is needed. Participants will be educated about signs of nicotine dependence and if they express interest in pharmacotherapy will be encouraged to access this through their personal healthcare providers. The Instagram groups will provide educational and social support, troubleshooting and advice about nicotine replacement therapy (NRT) or other forms of treatment.
  Interventions: Behavioral: Social Media Intervention
- Control Condition (No Intervention): Participants in the control condition will be directed to the Truth Initiative e-cigarette texting quit program. This innovative and free text message program was created with input from teens, college students and young adults who have attempted to, or successfully, quit e-cigarettes using text coaching methods

INTERVENTIONS:
Behavioral: Social Media Intervention — Social media based intervention using Instagram with up to 3 posts per day for 30 days
  Arms: Vaping Intervention

SUMMARY:
Social media based intervention to support teens in their efforts to quit vaping.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of a social media intervention to support teens in their efforts to quit vaping.

ELIGIBILITY:
Inclusion Criteria:

1. English literacy
2. Age between 13-21 years
3. Indicate they use social media "most" (>= 4) days per week
4. Have vaped at least once per week in the past 30 days (90 percent of participants)
5. Access to a computer or mobile phone with photo capability to verify abstinence from vaping
6. Indicate they are considering quitting or are interested in quitting with the next 6 months or within the next 30 days
7. Currently reside in California

Exclusion Criteria:

1. No English literacy
2. Age under 13 or over 21
3. Insufficient social media use (3 or fewer days per week)
4. Have not vaped at least once per week in past 30 days
5. No access to computer or mobile phone with photo capability to verify abstinence from vaping
6. Not considering or interested in quitting vaping in the next 30 days or 6 months;
7. Not a California resident

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Point Prevalent Abstinence (PPA) from vaping | 1 month
  7-day point prevalence abstinence (PPA) from all tobacco products will be assessed over the course of the study. Participants reporting no vaping in the past 7 days will be coded as abstinent. Those reporting 7-day abstinence and not using nicotine replacement therapy will be mailed saliva cotinine test kit and saliva tetrahydrocannabinol (THC) test kit for biochemical verification of abstinence.
Point Prevalent Abstinence (PPA) from vaping | 3 months
  7-day point prevalence abstinence (PPA) from all tobacco products will be assessed over the course of the study. Participants reporting no vaping in the past 7 days will be coded as abstinent. Those reporting 7-day abstinence and not using nicotine replacement therapy will be mailed saliva cotinine test kit and saliva tetrahydrocannabinol (THC) test kit for biochemical verification of abstinence.
Point Prevalent Abstinence (PPA) from vaping | 6 months
  7-day point prevalence abstinence (PPA) from all tobacco products will be assessed over the course of the study. Participants reporting no vaping in the past 7 days will be coded as abstinent. Those reporting 7-day abstinence and not using nicotine replacement therapy will be mailed saliva cotinine test kit and saliva tetrahydrocannabinol (THC) test kit for biochemical verification of abstinence.

SECONDARY OUTCOMES:
Change in the number of participants with reduction in vaping | Up to 6 months
  Reduction in vaping is defined as a decline in vaping frequency by 50 percent (%) or more.
Change in the number of vape quit attempts | Up to 6 months
  The number of quit attempts will be recorded at each assessment.
Number of participants with at least 1 quit attempt | Up to 6 months
  The number of participants whom achieved at least one quit attempt during the full assessment time period will be reported.
Change in response on Stages of Change Questionnaire | Up to 6 months
  The participants readiness to quit will be measured using the Stages of Change questionnaire - single item, which asks "Are you seriously thinking of quitting smoking?" Answers range from 'Yes, within the next 30 days', 'Yes, within the next 6 months', and 'No, not thinking of quitting'.
Change in the score on the Thoughts About Abstinence (TAA) Questionnaire | Up to 6 months
  The adapted Thoughts About Abstinence Questionnaire (Hall et al., 1991) is a 3 item self-report questionnaire that measures: 1) desire to quit smoking, 2) expected success at quitting, 3) expected difficulty of quitting on 10-point Likert scales (e.g., 1=no desire to quit/lowest expectation/lowest level of difficulty to 10 = extreme desire to quit/highest expectation of success/highest expected difficulty)
Change in the scores on the Ways of Quitting questionnaire (WOQ) | Up to 6 months
  The WOQ is a 28-item self-report instrument assessing adolescent smoking cessation strategies. For each WOQ item, respondents indicate whether they have used a given strategy (yes/no) and, if used, how helpful it was perceived to be on a five-point Likert-type scale (1= "Not helpful" to 5="Extremely helpful") with regard to several categories: Social support, Seeking assistance, Avoidance, Reduction, Substitution, Medication, Distraction, and Quit all at once (single item).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ling, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyu JC, Olson SS, Ramo DE, Ling PM. Delivering vaping cessation interventions to adolescents and young adults on Instagram: protocol for a randomized controlled trial. BMC Public Health. 2022 Dec 10;22(1):2311. doi: 10.1186/s12889-022-14606-7. PMID 36496358